CLINICAL TRIAL: NCT04491916
Title: A Cross-over Trial to Evaluate the Efficacy and Safety Between Increasing the Dose of Iron and Original Iron Dosage in Patients With Maintenance Hemodialysis
Brief Title: Iron Therapy in Patients With End-Stage Renal Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20190110
Record Dates: First submitted 2020-04-09; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2019-09

CONDITIONS: End-stage Renal Disease; Anemia; Cardiovascular Risk Factor; Inflammation
Keywords: iron; End-Stage Renal Disease; Anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Iron Treatment (Experimental): Treatment with iron sucrose with orginal guideline from ferritin>500ng/ml, or TSAT>20% to ferritin>800ng/ml, or TSAT>50%.
  Interventions: Drug: irone sucrose

INTERVENTIONS:
Drug: irone sucrose — drug ingredient: Ferric Hydroxide in complex with sucrose drug dosage form: 270injection/100mg/5ml/Amp

SUMMARY:
This study will compare the clinical outcome of patients with maintenance dialysis room after changing the iron treatment guidelines from original upper limit with ferritin>500ng/ml, or TSAT>20% to Ferritin> 800ng / ml, or TSAT> 50%.

DETAILED DESCRIPTION:
After two years of treatments, we will compare the incidence of clinical events, monthly blood, and biochemical examination data for the two years before and after the change.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving maintenance dialysis

Exclusion Criteria:

* less than 20 year-old, oncological patients undergoing chemotherapy, abnormal liver function, infection

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 2 years
  the death events following up until 2022
coronary artery disease | 2 years
  new onset coronary artery disease diagnosed with electrocardiogram (ST-segment changes, T inversion and Q wave appearance)
coronary artery disease | 2 years
  Progression of coronary artery disease (SCCT grading increase : 0% = no visible stenosis, 1-24% = minimal stenosis, 25-49% = mild stenosis, 50-69% = moderate stenosis, 70-99% = severe stenosis, 100% = occlusion)
coronary artery disease | 2 years
  new onset coronary artery disease diagnosed with cardiac enzyme (>troponins I upper limit 99%)
congestive heart failure | 2 years
  new onset congestive heart failure diagnosed with sonocardiogram (HF-REF, heart failure with reduced EF≦ 35%)
congestive heart failure | 2 years
  Progression of congestive heart failure (increase of NYHA classification)
congestive heart failure | 2 years
  new onset congestive heart failure with symptoms (Framingham's clinical criteria: orthopnea, pulmonary rales, S3, paroxysmal nocturnal dyspnea, cough, dyspnea on ordinary exertion, pleural effusion, hepatomegaly, tachycardia with a heart rate over 120 beats/min, bilateral leg edema, and weight loss under 4.5 kg in five days) diagnosed by cardiologists
congestive heart failure | 2 yearts
  new onset congestive heart failure (brain natriuretic peptide> 400pg/ml)

SECONDARY OUTCOMES:
diabetes | 2 years
  fasting blood sugar
diabetes | 2 years
  postprandial blood sugar
diabetes | 2 years
  glycated hemoglobin
anemia | 2 years
  1. serum hemoglobin level
  2. serum hematocrit
calcium | 2 years
  serum total calcium level
phospate | 2 years
  serum phosphate level
nutrition status | 2 years
  serum albumin level
liver function | 2 years
  serum AST/ALT level
liver function | 2 years
  abdominal sonography with Child classification of liver cirrhosis
sodium | 2 years
  serum sodium level
potassium | 2 years
  serum potassium level
parathyroid function | 2 years
  serum parathyroid level

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Y Lin, MD,PhD, Principal Investigator — Kaohsiung Medical University; Hugo Y Lin, MD,PhD, Principal Investigator — Kaohsiung Municipal Ta-Tung Hospital
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/16/NCT04491916/ICF_000.pdf